CLINICAL TRIAL: NCT04916392
Title: An Observational Study of the Pharmacokinetics of Adductor Canal Block Using Liposomal Bupivacaine and Standard Bupivacaine in Total Knee Arthroplasty Patients
Brief Title: Observation Study of the Pharmacokinetics of Adductor Canal Block
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Honorary Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW20-589
Record Dates: First submitted 2021-06-02; First posted 2021-06-07 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Toxicity, Drug
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liposomal bupivacaine: Nerve block will be preformed using 5ml of 1.33% liposomal bupivacaine with 5ml of 0.9% normal saline.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — 5ml of 1.33% liposomal bupivacaine with 5 ml of 0.9% normal saline will be given to treatment group.

SUMMARY:
With the aging of the population, osteoarthritis of knees and hips become major orthopedic problems worldwide. Osteoarthritis of the knees and hips is associated with a significant pain problem and functional disability. Total joints replacement is the ultimate surgical procedure to deal with such problems. Multimodal analgesia, including periarticular local infiltration of analgesia (LIA), regional nerve block using adductor canal block (ACB), opioid and non-opioid have been shown to be effective in managing postoperative pain. Regional nerve block using femoral nerve block or adductor canal block (ACB) is also a well-established analgesic technique after total knee replacement. Standard bupivacaine (SB), levobupivacaine, ropivacaine were used in ACB in these studies. Whether combining ACB with periarticular LIA has the additional benefit of prolonging analgesia or with synergistic effect remains controversial, because the number of RCTs conducted is not enough. Liposomal bupivacaine (LB) may further prolong the analgesic effect of ACB, as the therapeutic levels of bupivacaine are below the toxic range and sustained for 72 hours after injection. The purpose of this study is to evaluate the safety and systemic levels of serum bupivacaine following adductor canal block using LB 66.5mg in patients undergoing TKA with LIA over a 72-hour period. This also serves as a pilot study to determine the dose and timing of blood taking for serum bupivacaine level of a previously IRB approved study - "Comparing the efficacy of combining periarticular local infiltration of analgesia and adductor canal block using liposomal bupivacaine and standard bupivacaine- A prospective randomized controlled trial".

DETAILED DESCRIPTION:
After signing the consent form, participants will receive LIA with ACB using 5ml of 1.33% liposomal bupivacaine with 5ml of 0.9% normal saline.

Participants will receive routine preoperative, intraoperative, and postoperative treatments like other patients undergoing total knee replacement.

Blood will be collected during induction, at 1 hour, 2 hours, 4 hours, 8 hours, and 12 hours after the performance of ACB through a designated 14-gauge cannula, and also at 24, 48, and 72 hours after the operation during routine blood taking.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-80 years old
* Scheduled for elective primary unilateral total knee replacement
* Chinese patients
* BMI < 40
* Able to speak and understand Cantonese
* Able to provide informed oral and written consent

Exclusion Criteria:

* Single-stage bilateral total knee replacement
* Complex primary total knee replacement requiring the use of stem/augment/constrained liner
* Surgeries with significant intraoperative complications which may alter rehabilitation protocol e.g. collateral ligament injury, fracture requiring fixation
* Known allergy to opioids, local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2 inhibitors
* History of chronic pain other than chronic knee pain
* History of immunosuppression
* Daily use of glucocorticoids
* Daily use of strong opioids (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nicomorphine, oxycodone, or meperidine)
* History of severe heart disease (NYHA 2)
* Alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120 micromol/L
* Pre-existing neurological or muscular disorders
* Psychiatric illness or neurologic or psychiatric diseases potentially influencing pain perception
* Impaired or retarded mental state
* Difficulties in using patient-controlled analgesia (PCA)
* Pregnancy
* Local infection
* On immunosuppressants
* High BMI (>=40)
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for elective primary unilateral total knee replacement in Queen Mary Hospital.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Time to peak concentration of serum bupivacaine | 72 hours after the operation
  Serum bupivacaine will be quantified using High Performance Liquid Chromatography.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong